CLINICAL TRIAL: NCT06863142
Title: VRC 328: A Phase I Open-Label Clinical Trial to Evaluate the Dose, Safety, Tolerability, and Immunogenicity of Mosaic Hexavalent Influenza Vaccine VRC-FLUMOS0116-00-VP (FluMos-v2) With and Without ALFQ Adjuvant in Healthy Adults
Brief Title: Evaluating the Dose, Safety, Tolerability, and Immunogenicity of Mosaic Hexavalent Influenza Vaccine VRCFLUMOS0116-00-VP (FluMos-v2) With and Without ALFQ Adjuvant in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10002293; 002293-I
Record Dates: First submitted 2025-03-06; First posted 2025-03-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12-23

CONDITIONS: Influenza Prevention; Seasonal Influenza
Keywords: Dose - Escalation; Immune Response; Viral Infection; Respiratory Illness; Experimental Vaccine; Experimental Adjuvant; Influenza Vaccine
MeSH Terms: conditions — Virus Diseases; Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): 180 mcg of FluMos-v2 Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0116-00-VP
- Group 2 (Experimental): 60 mcg of FluMos-v2 + 0.5 ml of ALFQ Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0116-00-VP; Other: ALFQ
- Group 3A (Experimental): 180 mcg of FluMos-v2 + 0.5 ml of ALFQ Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0116-00-VP; Other: ALFQ
- Group 3B (Experimental): 180 mcg of FluMos-v2 + 0.5 ml of ALFQ Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0116-00-VP; Other: ALFQ

INTERVENTIONS:
Biological: VRC-FLUMOS0116-00-VP — The VRC-FLUMOS0116-00-VP (FluMos-v2) vaccine is composed of de novo engineered pentamer assembled with de novo engineered trimeric domains to an icosahedral core, projecting 20 HA ectodomain trimers from influenza strains: Influenza A (H1-H3) and Influenza B (Victoria lineage and Yamagata lineage)
Other: ALFQ — The ALFQ adjuvant is a sterile suspension that contains monophosphoryl 3-deacyl Lipid A [3D-PHAD(R)] and QS-21
  Arms: Group 2; Group 3A; Group 3B

SUMMARY:
Background:

Vaccines help the body learn to fight infections. Some vaccines are combined with adjuvants, which are added substances that make vaccines work better. FluMos-v2 is an experimental flu vaccine; ALFQ is an experimental adjuvant.

Objective:

To test FluMos-v2, with and without the ALFQ adjuvant, in healthy adults.

Eligibility:

Healthy adults aged 18 to 50 years. They must have received at least one flu vaccine from the 2020-21 season through the 2024-25 flu season. They must also agree not to receive the licensed 2025-26 flu vaccine.

Design:

Participants will have 12 clinic visits over 15 months.

Participants will be screened. They will have a physical exam and blood tests.

On 2 visits, about 4 months apart, participants will receive a vaccination. The shots will be given into the muscle of the upper arm. They will get a follow-up call the day after each shot. They will keep a daily diary for 7 days; they will record their temperature and any other symptoms they feel after each shot.

All clinic visits will include collection of blood, saliva, and nasal secretions. If participants develop flu symptoms (such as fever, runny nose, sore throat), they will be asked to come to the clinic.

About 2 weeks after each vaccination, participants may opt to undergo apheresis: Blood will be taken from the body through a needle inserted into one arm. The blood will pass through a machine that separates out the white blood cells. The remaining blood will be returned to the body through a needle in the other arm.

DETAILED DESCRIPTION:
Design:

This is a Phase I, open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of mosaic hexavalent influenza vaccine VRC-FLUMOS0116-00-VP (FluMos-v2) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) adjuvant. The hypotheses are that the FluMos-v2 vaccine is safe and tolerable when administered alone or with ALFQ adjuvant, that this vaccine elicits antigen-specific immune responses, and that addition of the ALFQ adjuvant increases the magnitude and breadth of the elicited immune responses. The primary objective is to evaluate the safety and tolerability of the investigational vaccine with and without ALFQ adjuvant in healthy adults. Secondary objectives are related to the immunogenicity of the investigational vaccine with and without ALFQ adjuvant.

Study Products:

The investigational vaccine FluMos-v2 was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID). The adjuvant, Army Liposome Formulation containing QS-21 (ALFQ), was developed, and provided by the Walter Reed Army Institute of Research (WRAIR).

The FluMos-v2 vaccine is composed of full-length HA trimers of the following 6 influenza strains:

Influenza A:

H1: A/Idaho/07/2018

H2: A/Singapore/1/1957

H3: A/Perth/1008/2019

H3: A/Darwin/106/2020

Influenza B:

B/Victoria lineage: B/Colorado/06/2017

B/Yamagata lineage: B/Phuket/3073/2013

VRC-FLUMOS0116-00-VP (FluMos-v2) is a sterile, aqueous buffered solution supplied in 3.0 mL single-dose glass vials containing 0.7 +/- 0.1 mL with a vaccine concentration of 180 mcg/mL.

The ALFQ drug product is a sterile suspension that contains 240 mcg of monophosphoryl 3-deacyl Lipid A (3D-PHAD(R)) and 120 mcg QS-21 that is vialed at 0.6 mL/vial in 3.0 mL glass vials. 0.5 mL of ALFQ adjuvant will be mixed with the 60 or 180 mcg dose of FluMos-v2 during preparation in the pharmacy prior to vaccination.

FluMos-v2 with and without ALFQ adjuvant will be administered intramuscularly (IM) in the deltoid muscle via needle and syringe.

Participants:

Healthy adults 18-50 years of age, inclusive, will be enrolled.

Study Plan:

Group 1 will open and enroll without any planned dose safety reviews, because the 180 mcg dose without adjuvant was evaluated as safe and tolerable in VRC 326 study. The adjuvanted dose groups, Groups 2, 3A, and 3B will proceed with the lower dose group enrolling first. There will be two interim dose safety reviews in this trial: the first will review the safety data for Group 2 (60 mcg of FluMos-v2 with ALFQ adjuvant). Enrollment for Group 2 will be limited to one participant per day for the first three participants. After the third participant's two-week post-vaccination visit, a safety review will decide whether to continue at the same dose level in Group 2 and open Group 3A and Group 3B to participants who will receive 180 mcg of FluMos-v2 with ALFQ adjuvant. Enrollment for Group 3A or Group 3B will also be limited to one participant per day for the first three participants. The second safety review is a dose continuation review for Group 3A and Group 3B (180 mcg of FluMos-v2 with ALFQ adjuvant). After the third participant's two-week post-vaccination visit, a safety review will determine whether to continue at the same dose level in Group 3A or Group 3B. Once all groups are open, participants will continue enrollment into each group at the discretion of the Principal Investigator (PI) to balance the number of enrollments in each group.

If a current participant is discontinued from the protocol, a new participant may be enrolled at the discretion of the PI in order to collect required safety or immunogenicity data.

Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

The study schema is as follows:

VRC 328 Vaccination Schema

Group - 1

Participants - 12

Day 0 - 180 mcg

Week 16 - 180 mcg

Product - FluMos-v2

Group - 2

Participants - 5

Day 0 - 60 mcg

Week 16 - 60 mcg

Product - FluMos-v2 + 0.5 mL ALFQ

Group - 3A

Participants - 12

Day 0 - 180 mcg

Week 16 - 180 mcg

Product - FluMos-v2 + 0.5 mL ALFQ

Group - 3B*

Participants - 0-6

Day 0 - 180 mcg

Week 16 - 180 mcg

Product - FluMos-v2 + 0.5 mL ALFQ

Total

Participants - 35**

*Enrollment in Group 3B is optional and includes participants who have previously taken part in the following influenza vaccine studies:

VRC 316 (ONLY participants enrolled in Groups 2, 3A, and 4A; HA-F A/Sing or DNA A/Sing vaccines) or VRC 321 (H1ssF_3928 vaccine) or VRC 323 (H10ssF-6473 vaccine).

**Enrollment of up to 45 participants is permitted if additional participants are needed for safety or immunogenicity evaluations.

Study Duration:

Participants will be evaluated for 68 weeks following the first vaccine administration, including through the 2025-2026 influenza season.

ELIGIBILITY:
* INCLUSION CRITERIA:
* A participant must meet all of the following criteria:

  * Healthy adults between the ages of 18-50 years, inclusive
  * Based on history and physical examination, be in good general health and without a history of any of the conditions listed in the exclusion criteria
  * Received at least one licensed influenza vaccine from the 2020-2021 influenza season through the 2024-2025 influenza season
  * Able and willing to complete the informed consent process
  * Available for clinic visits for 68 weeks after enrollment, including through the 2025-2026 influenza season
  * Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
  * Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) <= 35 within the 56 days before enrollment
  * Agrees to not receive the 2025-2026 licensed influenza vaccination during study participation due to potential confounding of study results
  * Willing to have blood and mucosal samples collected, stored indefinitely, and used for research purposes
* Laboratory Criteria within 56 days before enrollment

  * White blood cells (WBC) and differential within institutional normal range or accompanied by approval of the site Principal Investigator (PI) or designee
  * Total lymphocyte count >= 800 cells/microL
  * Platelets = 125,000 - 400,000 cells/microL
  * Hemoglobin within institutional normal range or accompanied by approval of the PI or designee
  * Alanine aminotransferase (ALT) <= 1.25 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) <= 1.25 x institutional ULN
  * Alkaline phosphatase (ALP) < 1.1 x institutional ULN
  * Total bilirubin within institutional normal range or accompanied by approval of the PI or designee
  * Serum creatinine <= 1.1 x institutional ULN
  * Negative for HIV infection by an FDA-approved method of detection
* Criteria applicable to women of childbearing potential:

  * Negative beta-human chorionic gonadotropin (Beta-HCG) pregnancy test (urine or serum) on the day of enrollment
  * Agrees to use an effective method of birth control from at least 21 days prior to enrollment through the end of the study.

EXCLUSION CRITERIA:

* A participant will be excluded if one or more of the following conditions apply:

  -- Women who are breast-feeding or planning to become pregnant during the study
* A Participant has received any of the following substances:

  * Receipt of any licensed influenza vaccine within 6 months prior to enrollment.
  * Plan to or are required to receive the 2025-2026 licensed influenza vaccine
  * Live attenuated vaccines within 4 weeks prior to enrollment
  * Inactivated vaccines within 2 weeks prior to enrollment
  * mRNA vaccines within 4 weeks prior to enrollment
  * Receipt of 20 mcg of the influenza vaccine VRC-FLUNPF081-00-VP (HA-F A/Sing, VRC 316, Group 1)
  * Receipt of the mosaic quadrivalent influenza vaccine VRC-FLUMOS0111-00-VP (FluMos-v1, VRC 325)
  * Receipt of the mosaic hexavalent influenza vaccine VRC-FLUMOS0116-00-VP (FluMos-v2, VRC 326)
  * More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
  * Blood products within 16 weeks prior to enrollment
  * Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
  * Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule
  * Current anti-TB prophylaxis or therapy
* Participant has a history of any of the following clinically significant conditions:

  * Serious reactions to vaccines that preclude receipt of the study vaccinations as determined by the PI or designee
  * Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
  * Asthma that is not well controlled
  * Diabetes mellitus (type I or II), except for gestational diabetes
  * Thyroid disease that is not well controlled
  * Idiopathic urticaria within the past year
  * Immune-mediated diseases, such as autoimmune or autoinflammatory diseases, or immunodeficiencies
  * Hypertension that is not well controlled
  * Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
  * Malignancy that is active or history of malignancy that is likely to recur during the period of the study
  * Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
  * Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
  * Guillain-Barre Syndrome
  * Any medical, social condition, occupational reason, or other reason that, in the judgment of the PI or designee, is a contraindication to protocol participation or impairs a participant s ability to give informed consent, including but not limited to clinically significant forms of infectious diseases, drug or alcohol abuse, autoimmune diseases, psychiatric disorders, or heart disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the FluMos-v2 (180 mcg) vaccine with ALFQ adjuvant administered to healthy adults at Day 0 and Week 16. | Through 68 weeks following the first vaccine administration, including through the 2025-2026 influenza season.
  To evaluate the safety and tolerability of a 2 dose regimen with ALFQ adjuvant.
Safety and tolerability of the FluMos-v2 (60 mcg) vaccine with ALFQ adjuvant administered to healthy adults at Day 0 and Week 16. | Through 68 weeks following the first vaccine administration, including through the 2025-2026 influenza season.
  To evaluate the safety and tolerability of a 2 dose regimen with ALFQ adjuvant.
Safety and tolerability of the FluMos-v2 (180 mcg) vaccine administered alone to healthy adults at Day 0 and Week 16. | Through 68 weeks following the first vaccine administration, including through the 2025-2026 influenza season
  To evaluate the safety and tolerability of a 2 dose regimen

SECONDARY OUTCOMES:
Antibody responses to the FluMos-v2 (180 mcg) vaccine administered alone as a 2 dose regimen to healthy adults at 2 weeks after each injection at Week 2 and Week 18. | Through 18 weeks following the first vaccine administration, including through the 2025-2026 influenza season.
  To evaluate antibody responses
Antibody responses to the FluMos-v2 (180 mcg) with ALFQ adjuvant vaccine administered as a 2 dose regimen to healthy adults at 2 weeks after each injection at Week 2 and Week 18. | Through 18 weeks following the first vaccine administration, including through the 2025-2026 influenza season.
  To evaluate antibody responses

CONTACTS AND LOCATIONS:
Overall Officials: Lasonji A Holman, C.R.N.P., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Widge AT, Hofstetter AR, Houser KV, Awan SF, Chen GL, Burgos Florez MC, Berkowitz NM, Mendoza F, Hendel CS, Holman LA, Gordon IJ, Apte P, Liang CJ, Gaudinski MR, Coates EE, Strom L, Wycuff D, Vazquez S, Stein JA, Gall JG, Adams WC, Carlton K, Gillespie RA, Creanga A, Crank MC, Andrews SF, Castro M, Serebryannyy LA, Narpala SR, Hatcher C, Lin BC, O'Connell S, Freyn AW, Rosado VC, Nachbagauer R, Palese P, Kanekiyo M, McDermott AB, Koup RA, Dropulic LK, Graham BS, Mascola JR, Ledgerwood JE; VRC 321 study team. An influenza hemagglutinin stem nanoparticle vaccine induces cross-group 1 neutralizing antibodies in healthy adults. Sci Transl Med. 2023 Apr 19;15(692):eade4790. doi: 10.1126/scitranslmed.ade4790. Epub 2023 Apr 19. PMID 37075129
- [Background] Ober Shepherd BL, Scott PT, Hutter JN, Lee C, McCauley MD, Guzman I, Bryant C, McGuire S, Kennedy J, Chen WH, Hajduczki A, Mdluli T, Valencia-Ruiz A, Amare MF, Matyas GR, Rao M, Rolland M, Mascola JR, De Rosa SC, McElrath MJ, Montefiori DC, Serebryannyy L, McDermott AB, Peel SA, Collins ND, Joyce MG, Robb ML, Michael NL, Vasan S, Modjarrad K; EID-030 Study Group. SARS-CoV-2 recombinant spike ferritin nanoparticle vaccine adjuvanted with Army Liposome Formulation containing monophosphoryl lipid A and QS-21: a phase 1, randomised, double-blind, placebo-controlled, first-in-human clinical trial. Lancet Microbe. 2024 Jun;5(6):e581-e593. doi: 10.1016/S2666-5247(23)00410-X. Epub 2024 May 15. PMID 38761816
- [Background] Boyoglu-Barnum S, Ellis D, Gillespie RA, Hutchinson GB, Park YJ, Moin SM, Acton OJ, Ravichandran R, Murphy M, Pettie D, Matheson N, Carter L, Creanga A, Watson MJ, Kephart S, Ataca S, Vaile JR, Ueda G, Crank MC, Stewart L, Lee KK, Guttman M, Baker D, Mascola JR, Veesler D, Graham BS, King NP, Kanekiyo M. Quadrivalent influenza nanoparticle vaccines induce broad protection. Nature. 2021 Apr;592(7855):623-628. doi: 10.1038/s41586-021-03365-x. Epub 2021 Mar 24. PMID 33762730
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002293-I.html